CLINICAL TRIAL: NCT00289861
Title: Risperidone Augmentation in Patients With Schizophrenia Partially Responsive to Clozapine
Brief Title: Risperidone Augmentation in Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Oliver Freudenreich, Medical Director, MGH Schizophrenia Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2002-P-000584
Record Dates: First submitted 2006-02-08; First posted 2006-02-10 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; risperidone; prolactin; clozapine
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- risperdone (Active Comparator)
  Interventions: Drug: Risperidone
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Risperidone
  Arms: risperdone
Drug: placebo
  Arms: placebo

SUMMARY:
We propose a double-blind, placebo-controlled trial to study the effectiveness and tolerability of adding risperidone to stable yet only partially remitted patients with schizophrenia maintained on clozapine.

DETAILED DESCRIPTION:
Specific Aims - We propose a double-blind, placebo-controlled trial to study the effectiveness and tolerability of adding risperidone to stable yet only partially remitted patients with schizophrenia maintained on clozapine. We anticipate enrolling a total of 40 subjects over a period of two years at the Freedom Trail Clinic and affiliated sites in Boston, Massachusetts. Our primary outcome measure will be change in total score on the Positive and Negative Syndrome Scale (PANSS). Secondary hypotheses are (1) that the clozapine-risperidone combination is well tolerated, (2) that clozapine levels will not be influenced by risperidone, and (3) that prolactin elevation is suitable as a surrogate marker of sufficient D2 blockade to predict response.

Background - Despite a new generation of antipsychotics, many patients with schizophrenia achieve only partial syndromal remission. In an effort to improve symptomatic and functional outcomes, it has become common practice to combine antipsychotic medications. Since this strategy is largely unproven and expensive, empirical trials are urgently needed. Our group has found in an open trial that adding risperidone to clozapine was well tolerated and led to improvement in psychopathology. Additional support for increasing D2 blockade in clozapine partial responders comes form two small studies using sulpiride and pimozide. We hypothesize that there is a subgroup of patients who might benefit from additional D2 blockade beyond what clozapine alone accomplishes.

Methods - The proposed trial will be placebo-controlled, randomized, and double-blind, and it will last 8 weeks. We expect to enroll 40 subjects overall. Subjects will be eligible if they are diagnosed with schizophrenia and treated with clozapine. In addition, they must have residual symptoms of schizophrenia as we are interested in improvement of residual psychopathology. Subjects with dementia or mental retardation as well as pregnant women will be excluded. After a 2-week placebo lead-in period to assure stable psychopathology and minimize placebo-response, subjects will be randomly allocated to receive 6 weeks of either risperidone (20 subjects), or matching placebo (20 subjects) added onto their customary antipsychotic medication, clozapine. Overall, there are 5 study visits every 2 weeks plus the initial screening visit. On each visit, subjects will be evaluated with standard psychiatric rating scales of psychopathology and side effects. In addition, we will measure serum levels of the medications used, clozapine and risperidone.

Fasting glucose will be measured at screening, week 4, and week 8 visits. This is done to monitor subjects for worsening glucose control. This is a possible concern due to the association between atypical antipsychotics, including risperidone, and hyperglycemia. Subjects who are discovered to either have diabetes or develop diabetes during the study, or who have worsening glucose control if diabetic, will be discontinued and referred to their PCP for further work-up and treatment. This additional blood test will not lead to additional blood draws but will simply be added to the subject's routine and mandated biweekly WBC monitoring.

The study endpoint will be a 20% improvement on our primary rating scale of psychopathology, the Positive and Negative Syndrome Scale (PANSS). No worsening of psychopathology is expected in this trial as subjects are maintained on primary antipsychotic, clozapine.

Benefits - There are no definite benefits to participating in this trial. Subjects will receive a thorough psychiatric evaluation, a review of their pharmacologic treatment, and a physical exam with some baseline laboratory studies. The results of the initial evaluation will be communicated to the treating psychiatrist. Subjects will receive a nominal fee of $20 per study visit (5 study visits are scheduled overall).

The proposed study has direct clinical applications, and it is of theoretical interest. Few data are available from controlled trials to guide clinicians when patients remain symptomatic on clozapine. From a conceptual standpoint, the study will clarify the value of additional D2 blockade for treatment response.

Risks and Discomforts - Risperidone is approved by the FDA for the treatment of schizophrenia. The dose of 4 mg is on the lower end of the dosing recommendations and is usually well tolerated. Possible side effects are sedation, extrapyramidal symptoms, akathisia, hyperprolactinemia, or orthostatic hypotension. Tardive dyskinesia is a long-term side effect and would not be expected in a 6-week trial. However, existing tardive dyskinesia could worsen.

Blood drawing entails transient discomfort, and it might lead to a hematoma at the site. Being interviewed for clinical symptoms with the help of rating scales can be tiring and upsetting if sensitive psychological experiences are discussed. There is also an association between atypical antipsychotics, including risperidone, and hyperglycemia, requiring some monitoring of blood sugars during treatment. No inpatient hospital time is required.

Minimization of Risks - To minimized discomfort from blood draws, the study blood work will be added onto the mandatory blood draws that subjects undergo because they receive clozapine. Vital signs will be monitored at baseline and every two weeks. Side effects will be monitored at baseline and every two weeks. The Systematic Assessment for Treatment Emergent Events (SAFTEE) will be the primary instrument used to detect side effects. The SAFTEE will be used to tabulate side effects for the yearly IRB summary. Serious adverse events, as well as adverse events, will be reviewed by the PI and reported to the IRB according to institutional policy. The PIs in our group meet weekly to review study protocols and study events.

Fasting glucose will be measured at screening, week 4, and week 8 visits. This is done to monitor subjects for worsening glucose control. This is a possible concern due to the association between atypical antipsychotics, including risperidone, and hyperglycemia. Subjects who are discovered to either have diabetes or develop diabetes during the study or who have worsening glucose control (poor glucose control as judged by new-onset diabetes or new-onset glucose intolerance.) will be discontinued and referred to their primary care physician (PCP) for further work-up and treatment. In patients with established diabetes, the six weeks of active treatment will not be long enough to meaningfully judge if diabetes control is more difficult than usual (typical parameters of glucose control such as hemoglobin A1C are a reflection of long-term glucose control, i.e. several months). We will follow those patients clinically in cooperation with the PCP to decide if patients can stay in the trial. This additional blood test will not lead to additional blood draws but will simply be added to the subject's routine and mandated biweekly white blood cell count monitoring.

Patients will be withdrawn from the study if they become suicidal or deteriorate psychiatrically. This will be assessed every 2 weeks using the PANSS and Calgary Depression Scale for Schizophrenia (CDSS): clinical deterioration will be defined as a 20% increase in total PANSS scores, and suicidality will be defined as a rating of "mild" (frequent thoughts of being better off dead, or occasional thought of suicide) on the CDSS. Subjects who have worsening symptoms of tardive dyskinesia (TD) will be discontinued and referred to their psychiatrist for further work-up and treatment (Worsening TD as judged by 20% increase in Abnormal Involuntary Movement Scale (AIMS)).

ELIGIBILITY:
Inclusion Criteria:

1. Clinical DSM-IV diagnosis of schizophrenia (any subtype) based on chart review and patient interview by research psychiatrist
2. Ages 18-65
3. Stable residual psychiatric symptoms defined as PANSS score greater than 60
4. On clozapine monotherapy with plasma level of at least 200 ng/mL (unless the patient refuses a dose adjustment or does not tolerate a higher dose)
5. On clozapine for at least 6 months and at a stable dose for at least 8 weeks
6. Competent to provide informed consent. If the subject has a guardian, assent must be given by the subject and consent must be given by the guardian.

Exclusion Criteria:

1. Chart diagnosis of dementia or another neurodegenerative disorder, mental retardation, or a pervasive developmental disorder
2. Suicidal ideation
3. Substance use disorder (excluding nicotine use) in the past 3 months
4. Any unstable medical illness
5. Pregnancy or breast-feeding
6. Investigational agent in past 30 days
7. History of adverse reaction to risperidone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Our primary outcome measure will be change in total score on the Positive and Negative Symptom Scale (PANSS).

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Freudenreich, M.D., Principal Investigator — MGH; Donald C Goff, M.D., Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Freudenreich O, Henderson DC, Walsh JP, Culhane MA, Goff DC. Risperidone augmentation for schizophrenia partially responsive to clozapine: a double-blind, placebo-controlled trial. Schizophr Res. 2007 May;92(1-3):90-4. doi: 10.1016/j.schres.2006.12.030. Epub 2007 Feb 23. PMID 17321111